CLINICAL TRIAL: NCT06575907
Title: Health, Functioning, Work, and Experiences of Social and Health Services of Persons With Stroke
Acronym: FinPostStroke
Status: Active, not recruiting | Type: Observational
Sponsor: The Finnish Association of People with Physical Disabilities (Other)
Collaborators: HUS Helsinki University Hospital (Unknown); Kuopio University Hospital (Other); The Finnish Brain Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: pr42115
Record Dates: First submitted 2024-08-21; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Stroke; Health, Subjective; Cardiovascular Diseases; Central Nervous System Diseases
Keywords: ICF; Survey; Stroke; Health; Functioning; Work; Inclusion; Health and social services
MeSH Terms: conditions — Stroke; Cardiovascular Diseases; Central Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Persons treated in Kuopio University Hospital
  Interventions: Other: no intervention
- Persons treated in HUS Helsinki University Hospital
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The purpose of the Health, functioning, work, and experiences of social and health services of persons with stroke study (FinPostStroke) is to identify factors related to self-reported health, functioning, work, inclusion, and accessibility of social and health services, and how such factors are interconnected in Finnish adults one or more years after stroke. Participants will be targeted from two tertiary hospitals' registries and recruited via mail.

This cross-sectional explorative observational study is based on register data and postal survey. The survey questionnaire includes several valid patient-reported outcome measures. The study will add knowledge to be utilized in developing health care and rehabilitation services for people with stroke, as well as provide information for various parties involved.

DETAILED DESCRIPTION:
The purpose of the Health, functioning, work, and experiences of social and health services of persons with stroke (FinPostStroke) study is to identify factors related to self-reported health, functioning, work, inclusion, and accessibility of social and health services, and how such factors are interconnected in Finnish adults one or more years after stroke. The International Classification of Functioning, Disability and Health (ICF) is used as a structured framework.

Adults with cerebral infarction, subarachnoid hemorrhage, or intracerebral hemorrhage will be targeted from Kuopio and HUS Helsinki University Hospitals' patient registries. The survey data is planned to be collected with postal questionnaire by May 2025. The questionnaire includes several valid patient-reported outcome measures to assess health and functioning, work and income, inclusion, and social and health services. Participants will be recruited via mail with an invitation letter and study information attached to the questionnaire. All participants are expected to give written informed consent prior to the study.

This study will add knowledge to be utilized in developing health care and rehabilitation services for people with stroke, as well as provide information for various parties involved. We plan to publish at least four peer-reviewed articles along with common articles and texts concerning self-reported health, functioning, work, inclusion, and accessibility of social and health services among Finnish adults with stroke.

ELIGIBILITY:
Inclusion Criteria:

* treated for a stroke (ICD-10 codes I60-61, I63-64) in HUS Helsinki University Hospital or in Kuopio University Hospital between January 2018 and December 2022
* stroke is primary diagnose for the treatment
* 18 years or older at the time of survey

Exclusion Criteria:

* stroke is secondary diagnose for the treatment
* treated for a stroke only as outpatient in other than emergency room
* lives abroad
* missing address

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with cerebral infarction, subarachnoid hemorrhage, or intracerebral hemorrhage that have been treated either in Kuopio or HUS Helsinki University Hospitals in 2018-2022.
Sampling Method: Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
PROMIS® Global Health | 7 days
  The Patient-Reported Outcomes Measurement Information System (PROMIS®) General Health consists of 10 items with 5-point rating scale. It is used to assess overall health, physical health, mental health, social health, fatigue, and pain.
PROMIS® 29+2 Profile | 7 days
  The Patient-Reported Outcomes Measurement Information System (PROMIS®) 29+2 Profile consists of 31 items with 5-point rating scale. It is used to assess physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference and intensity, and cognitive function.
12-item WHODAS 2.0 | 30 days
  The 12-item World Health Organization Disability Schedule 2.0 (WHODAS) measures functioning. It consists of 12 items with 5-point rating scale (0-4), sum score ranging from 0 to 48. Higher score means more disability. It is used to assess cognition, mobility, self-care, getting along, life activities, and participation.
Experiences of Social Inclusion Scale, ESIS | 1 day
  Experiences of Social Inclusion Scale (ESIS) consists of 10 claims with 5-point Likert scale (1-5). The sum score of 10-50 is converted to a scale of 0 to 100. Higher score means stronger experience of inclusion. It is used to assess the experience of meaningfulness, belief in action possibilities and the perceived quality of social interaction.
Health and social services | 1 year
  "Health and social services" consists of 24 semistructured questions about health and social services chosen from the National Health Finland Survey.
Work and income | 30 days
  "Work and income" consists of 14 semistructured questions about work and income chosen from the International Spinal Cord Injury Survey.

CONTACTS AND LOCATIONS:
Overall Officials: Sinikka Hiekkala, Principal Investigator — The Finnish Association of People with Physical Disabilities
Locations (1):
- The Finnish Association of People with Physical Disabilities, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No